CLINICAL TRIAL: NCT00768027
Title: Outcome Assessment in Patients Treated With Hyperbaric Oxygen Using OxyVu Tissue Oxygenation Monitoring System
Acronym: HBOT
Status: Suspended | Type: Observational
Why Stopped: Seeking additional funds
Sponsor: HyperMed (Industry)
Collaborators: Hyperbaric and Wound Care Associates (Unknown); VA Long Beach Healthcare System (U.S. Federal Agency); Long Beach Memorial Medical Center (Other)
Responsible Party: Kevin Schomacker, PhD, HyperMed, Inc.
Other Study IDs: 2008-012
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Wounds
Keywords: hyperspectral imaging; tissue oxygenation; wounds; wound healing; prevention; hyperbaric
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective is to define patient eligibility for hyperbaric oxygen therapy and to evaluate wound healing progression using a new hyperspectral imaging technology.

DETAILED DESCRIPTION:
The purpose of this clinical study is to define patient eligibility for hyperbaric oxygen therapy (HBOT) and to evaluate wound healing progression during HBOT using a new hyperspectral imaging technology (OxyVu).

ELIGIBILITY:
Inclusion criteria:

* 18 - 85 years of age
* Patients with wounds that meet the criteria for hyperbaric oxygen therapy (e.g. problem wound, diabetic foot ulcer, necrotizing soft tissue infections)
* Compromised Flap or Grafts.

Exclusion criteria:

* Patients with poor cardiac output (EF < 20%)
* Patients with severe obstructive pulmonary disease who don't qualify for HBOT
* Patients with untreated asthma who don't qualify for HBOT
* Patients utilizing supplemental oxygen and those on ventilators
* Patients on life support medications (pressors)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 to 85 years of age, males and females, and with and without diabetes and untreatable peripheral vascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
OxyVu measurements will be compared to transcutaneous oxygen measurements pre and post HBOT | Days 1, 7, 14, 21, 4wks, and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Niezgoda, MD, Principal Investigator — Hyperbaric & Wound Care Associates; Ian L Gordon, MD PhD, Principal Investigator — VA Long Beach Healthcare System; Michael B Strauss, MD, Principal Investigator — Long Beach Memorial Medical Center
Locations (3):
- United States (3):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Long Beach VA Medical Center, Long Beach, California
  - Hyperbaric & Wound Care Associates, Milwaukee, Wisconsin

REFERENCES:
- [Background] Mathieu D. Role of hyperbaric oxygen therapy in the management of lower extremity wounds. Int J Low Extrem Wounds. 2006 Dec;5(4):233-5. doi: 10.1177/1534734606294450. No abstract available. PMID 17088598
- [Background] Niinikoski JH. Clinical hyperbaric oxygen therapy, wound perfusion, and transcutaneous oximetry. World J Surg. 2004 Mar;28(3):307-11. doi: 10.1007/s00268-003-7401-1. Epub 2004 Feb 17. PMID 14961187
- [Background] Niinikoski J. Hyperbaric oxygen therapy of diabetic foot ulcers, transcutaneous oxymetry in clinical decision making. Wound Repair Regen. 2003 Nov-Dec;11(6):458-61. doi: 10.1046/j.1524-475x.2003.11610.x. PMID 14617286
- [Background] Fife CE, Buyukcakir C, Otto GH, Sheffield PJ, Warriner RA, Love TL, Mader J. The predictive value of transcutaneous oxygen tension measurement in diabetic lower extremity ulcers treated with hyperbaric oxygen therapy: a retrospective analysis of 1,144 patients. Wound Repair Regen. 2002 Jul-Aug;10(4):198-207. doi: 10.1046/j.1524-475x.2002.10402.x. PMID 12191001
- [Background] Fife CE, Buyukcakir C, Otto G, Sheffield P, Love T, Warriner R 3rd. Factors influencing the outcome of lower-extremity diabetic ulcers treated with hyperbaric oxygen therapy. Wound Repair Regen. 2007 May-Jun;15(3):322-31. doi: 10.1111/j.1524-475X.2007.00234.x. PMID 17537119
- [Background] Niezgoda JA, Mewissen M. The management of lower extremity wounds complicated by acute arterial insufficiency and ischemia. Ostomy Wound Manage. 2004 May;50(5A Suppl):1-11; quiz 12. PMID 15366447
- [Background] Deerochanawong C, Home PD, Alberti KG. A survey of lower limb amputation in diabetic patients. Diabet Med. 1992 Dec;9(10):942-6. doi: 10.1111/j.1464-5491.1992.tb01736.x. PMID 1478041
- [Background] Frykberg RG. Guidelines for diabetic foot care. Foot Ankle Int. 2000 Jul;21(7):616. doi: 10.1177/107110070002100716. No abstract available. PMID 10919631
- See also: Sponsor and OxyVu technology website — http://www.hypermed-inc.com